CLINICAL TRIAL: NCT05188664
Title: A Phase I/II, Open-Label, Multiple Centre Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM- 302 in Combination With Toripalimab in Patients With Advanced Solid Tumors
Brief Title: Study of LaNova Medicines(LM)-302 in Combination With Toripalimab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Australia Pty Limited (Industry)
Responsible Party: Sponsor
Organization: LaNova Medicines Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM302-01-201
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: This study includes two stages, Phase I (Dose escalation) which includes LM-302 monotherapy dose escalation (part Ia) and LM-302 in combination with Toripalimab therapy dose escalation (part Ib) and Phase II (Dose expansion).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LM-302 monotherapy dose escalation (Experimental): LM-302 monotherapy dose escalation (part Ia). Accelerated titration combined with traditional 3+3 design will be used for monotherapy dose escalation (part Ia).
  Interventions: Drug: LM-302
- LM-302 in combination therapy dose escalation (Experimental): LM-302 in combination therapy dose escalation (part Ib).Accelerated titration combined with traditional 3+3 design will be used for LM-302 in combination with fixed dose Toripalimab dose escalation (part Ib).
  Interventions: Drug: LM-302; Drug: Toripalimab
- LM-302 Dose Expansion (Experimental): SMC will select appropriate dose(s) and/or tumor types for dose expansion study.
  Interventions: Drug: LM-302; Drug: Toripalimab

INTERVENTIONS:
Drug: LM-302 — LM-302 is given by intravenous (IV) infusion on day 1 every 3 weeks。
Drug: Toripalimab — Toripalimab with a fixed dose is given by intravenous (IV) infusion on day 1 every 3 weeks.
  Other Names: Tuoyi
  Arms: LM-302 Dose Expansion; LM-302 in combination therapy dose escalation

SUMMARY:
A Phase I/II, Open-Label, Multiple Centre Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM- 302 in Combination with Toripalimab in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a study of LM-302 in combination with toripalimab in patients with advanced solid tumors .The study includes phase I (dose escalation) and phase II (dose expansion). All participants enrolled in the study will be administered every 3 weeks (1 cycle=21 days) with a dose of LM-302 intravenous infusion followed by toripalimab intravenous infusion on day 1 until meet the criteria of treatment discontinuation or withdraw, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged ≥18 years old when sign the ICF, male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, and no deterioration within 2 weeks prior to the first dose.
4. Life expectancy ≥ 3 months.
5. Subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumors, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
6. CLDN18.2 test should be performed for the enrolled subjects if the archived tumor tissue samples are available.
7. At least one measurable lesion for phase II dose expansion, according to RECIST v1.1 as assessed by the investigator.
8. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose:

   1. Bone marrow reserve: Platelet count (PLT) ≥ 90 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Haemoglobin ≥ 9 g/dL, without receiving EPO, G-CSF, or GM-CSF within 14 days and blood transfusion including red blood cell and platelet transfusion in at least 7 days prior to first dose.
   2. Coagulation function: INR ≤ 1.5; APTT ≤ 1.5 × ULN.
   3. Liver function: Total bilirubin ≤ 1.5 × ULN (Subjects with Gilbert's Syndrome are allowed if total bilirubin ≤ 3 × ULN); AST and ALT ≤ 2.5 × ULN without liver metastases (≤ 5 × ULN if liver metastases are present); Albumin ≥ 2.5 g/dL.
   4. Kidney function: Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min.
   5. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; QT interval (QTcF) ≤ 480 ms.
9. Subjects who are able to communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Participate in any other clinical trial within 28 days prior to 1st dosing of investigational medicinal product (IMP).
2. Subjects with anti-tumor treatment within 21 days prior to 1st dosing of IMP, including radiotherapy, chemotherapy, biotherapy, endocrine therapy and immunotherapy, etc. the following treatments have different time limits:

   1. Local small-scale palliative radiotherapy (bone metastasis radiotherapy to control pain) within 14 days prior to 1st dosing.
   2. Oral anti-tumor therapy, including fluorouracil antitumor drugs and small molecular targeted drugs, etc. within 14 days or 5 half-lives of the drug (whichever is longer) prior to 1st dosing.
   3. Traditional herbal medicine with anti-tumor indication within 14 days prior to 1st dosing.
   4. Nitrosourea or Mitomycin C within 42 days prior to 1st dosing.
3. Subjects who experienced grade 3 or higher hypersensitivity to the treatment that contains monoclonal antibody, e.g., monoclonal antibody therapy, ADC etc.
4. Subjects who were intolerable to the treatment with MMAE based ADCs or anti-CLDN18.2 antibodies, but they can be enrolled if they were tolerable to the treatments and have experienced a 28-day's washout period prior to 1st dosing of IMP.
5. Subjects who were intolerable to the immunotherapy targeting PD-1 receptor, or its ligand PD-L1.
6. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
7. Administrate strong inhibitors/strong inducers of CYP3A4 within 14 days prior to 1st dosing of IMP.
8. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications.
9. Pre-existing peripheral sensory or motor neuropathy ≥ Grade 2.
10. Subjects with uncontrolled pain. Subjects requiring analgesic treatment must be on a stable regimen before participating in the study.
11. Subjects with known central nervous system (CNS) or meningeal metastasis.
12. Subjects who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
13. Subjects with known active keratitis or corneal ulcerations.
14. Use of any live attenuated vaccines within 28 days prior to 1st dosing of IMP.
15. Subjects with the history of idiopathic pulmonary fibrosis, organizing pneumonia.
16. Subjects with the known history of autoimmune disease.
17. Subjects who are taking therapeutic doses of anticoagulants.
18. Subjects with gastric outlet obstruction, persistent recurrent vomiting or uncontrolled/severe gastrointestinal hemorrhage, or ulcer within 28 days prior to 1st dosing of IMP.
19. Subjects who received major surgery or interventional treatment within 28 days prior to 1st dosing of IMP.
20. Subjects who have other active malignancies which are likely to require the treatment.
21. Subjects who have severe cardiovascular disease.
22. Subjects who have uncontrolled or severe illness, including but not limited to ongoing or active infection (e.g., active COVID-19/SARS-CoV-2 infection, etc.) requiring therapeutic antibiotics and/or other administration, while SARS-CoV-2 testing is not mandatory for study entry, and the testing should follow local clinical practice guidelines/standards.
23. Subjects who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation, or allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation.
24. HIV infection, active HBV and HCV infection.
25. Child-bearing potential female who have positive results in pregnancy test or are lactating.
26. Subjects who have psychiatric illness or disorders that may preclude study compliance; Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
DLT | Cycle 1 of each cohort. Duration of one cycle is 21 days
  To assess the safety and tolerability for LM-302 in combination with toripalimab in subjects with advanced solid tumors.
RP2D | Up to 6 months
  Obtain the recommended phase 2 dose (RP2D) for LM-302 in combination with toripalimab in subjects with advanced solid tumors.
OBD | Up to 6 months
  Obtain the optimal biologic dose (OBD) for LM-302 in combination with toripalimab in subjects with advanced solid tumors.
MTD | Up to 21 days
  Obtain the Maximum Tolerated Dose (MTD) for LM-302 in combination with toripalimab in subjects with advanced solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Ganju, Principal Investigator — Peninsula & South Eastern Haematology and Oncology Group; Ben Markman, Principal Investigator — The Alfred; Sophia Frentzas, Principal Investigator — Monash Medical Centre Clayton; Sara Wahlroos, Principal Investigator — Chris O'Brien Lifehouse; Jessica Smith, Principal Investigator — Macquarie University
Locations (1):
- The Alfred, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No